CLINICAL TRIAL: NCT06258044
Title: The Application Value of Deep Learning-Based Nomograms in Benign-Malignant Discrimination of TI-RADS Category 4 Thyroid Nodules
Status: Completed | Type: Observational
Sponsor: Ma Zhe (Other)
Responsible Party: Sponsor-Investigator, Ma Zhe, Director of Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(133)
Record Dates: First submitted 2024-01-04; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Nodule
Keywords: TI-RADS category 4 thyroid nodules; YOLOv3 model; nomograms
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- maligant: Thyroid nodules with surgical or puncture biopsy-confirmed pathological findings of malignancy in the TI-RADS4 category
- benign: Thyroid nodules with surgical or puncture biopsy-confirmed pathological findings of benign TI-RADS4 category

SUMMARY:
This retrospective study focuses on benign and malignant classification of thyroid nodules using deep learning techniques and evaluates the value of deep learning based nomograms in the classification of TI-RADS category 4 thyroid nodules to improve the accuracy of benign and malignant identification of TI-RADS category 4 thyroid nodules.

Materials and methods: Patients who visited in The First Affiliated Hospital of Shandong First Medical University ＆ Shandong Provincial Qianfoshan Hospital were collected. Their general clinical features, information on preoperative ultrasound diagnosis, and postoperative pathologic data were reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Ultrasound-confirmed diagnosis of thyroid nodules that are classified as TI-RADS category 4.
2. Availability of pathological results.

Exclusion Criteria:

1. Lack of pathological diagnosis.
2. History of thyroid surgery or other treatments.
3. Poor quality of ultrasound images of thyroid nodules.
4. Incomplete clinical and imaging data of the patient.

Ages: 23 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study collected data on a total of 500 TI-RADS category 4 thyroid nodules from 500 patients who attended the First Affiliated Hospital of Shandong First Medical University from April 2022 to November 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
deep learning prediction model（YOLOv3） and the model evaluation | Immediately evaluated after the prediction model was built
  Based on the characteristics of benign and malignant thyroid nodules, the dataset was divided into a training set and a test set using the cross-validation method, and the YOLOv3 model was trained using data from the training set, and the performance of the model was evaluated using data from the test set.The model is evaluated using a number of metrics such as: precision-recall curve, effective classification precision, confusion matrix and area under the curve.
nomogram prediction and assessment | Immediately evaluated after the nomogram was built
  Factoring clinical features, ultrasound grading and model predictions to map nomograms using R language.Evaluation of the nomogram using various metrics, including subject operating characteristic curves, calibration curves and decision curve analysis
Selection of clinical features and assessment | After the dataset is collected and pathology results are obtained, the statistical results obtained are analyzed for clinical factors, averaging about 1 year.
  The researchers selected patients with TI-RADS category 4 thyroid nodules within 1 year to comprise the dataset. The researchers analyzed the clinical factors in the dataset and analyzed the significance of these clinical factors on the statistical results and clinical characteristics using the Wilcoxon two-sample rank sum test or chi-square test.
Impact and assessment of ultrasound grading | The graded results of the ultrasound examination were analyzed after the data set collection was completed, the ultrasound examination was completed and the final pathology results were obtained, on average about 1 year.
  The researchers selected patients with TI-RADS category 4 thyroid nodules within 1 year to comprise the dataset. The researchers analyzed the results of grading TI-RADS category 4 nodules in this dataset and determined the significance of ultrasound grading on the statistical results using the chi-square test.

CONTACTS AND LOCATIONS:
Locations (1):
- QianfoshanH, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No